CLINICAL TRIAL: NCT06020066
Title: Stereotactic Radiotherapy for Non-small Cell Lung Cancer With Oligo-residual Intracranial Disease After First-line Third-generation EGFR Inhibitors: a Multicenter, Randomized Clinical Trial.
Brief Title: SRS for NSCLC With Oligo-residual Intracranial Disease After First-line 3rd Generation EGFR-TKI
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhengfei Zhu, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2306276-14
Record Dates: First submitted 2023-08-18; First posted 2023-08-31 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Brain Metastases; Non-small Cell Lung Cancer
MeSH Terms: conditions — Brain Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 3rd generation EGFR-TKI+SRS (Experimental): The experimental arm will undergo stereotactic radiotherapy targeting all residual lesions in the brain (completed in a single or multiple treatment courses within one month), while continuing EGFR-TKI therapy until disease progression or intolerable toxicity occurs.
  Interventions: Drug: EGFR-TK Inhibitor; Radiation: Stereotactic radiotherapy
- 3rd generation EGFR-TKI (Active Comparator): The control group will receive 3rd generation EGFR-TKI until disease progression or intolerable toxicity occurs.
  Interventions: Drug: EGFR-TK Inhibitor

INTERVENTIONS:
Drug: EGFR-TK Inhibitor — Patients will receive EGFR-TKI until confirmed progression or unacceptable toxicity.
Radiation: Stereotactic radiotherapy — Patients with oligo-residual intracranial disease after treatment with EGFR-TKI will be treated with SRS of all intracranial lesions. The choice of dose-fractionation regimen is at the discretion of the treating radiation oncologist.
  Arms: 3rd generation EGFR-TKI+SRS

SUMMARY:
Despite the impressive response rate to third-generation EGFR-TKIs, resistance inevitably develops in most patients. Stereotactic radiotherapy plays a growing role in the management of patients with brain metastasis. This study aims to evaluate the efficacy and safety of stereotactic radiotherapy for oligo-residual intracranial disease after first-line third-generation EGFR Inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed non-small cell lung cancer;
* Clinical stage IV (AJCC, 8th edition, 2017);
* EGFR mutations: EGFR L858R, EGFR exon 19 deletion;
* Age ≥18 years;
* KPS score ≥70;
* Brain metastasis at the time of diagnosis;
* Complete baseline imaging assessment of metastatic lesions, including enhanced MRI for brain;
* Receiving first-line treatment with third-generation EGFR inhibitors;
* After 3-6 months of third-generation EGFR inhibitor treatment, imaging review indicates no progression of extracranial lesions, and brain lesions are evaluated by thin-layer (1mm layer) enhanced MRI, meeting the following criteria:

  * No more than 10 remaining brain lesions;

    * The maximum diameter of the remaining brain lesions does not exceed 3cm;

      * At least one remaining brain lesion has a diameter greater than 5mm;

        * After evaluation by the researcher, all remaining brain lesions are suitable for stereotactic radiotherapy.
* Patient informed consent.

Exclusion Criteria:

* Poor compliance with the study protocol in the investigator's opinion;
* Patients withdrew their informed consent and requested to withdraw from the study;
* Patients were unable to receive regular doses of third-generation EGFR inhibitors due to other underlying conditions, viral side effects, economic factors, etc. (e.g., continuous discontinuation for more than 1 week, cumulative discontinuation for more than 2 weeks).
* Patients did not follow the protocol for follow-up visits as required by this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2027-08-10 (Estimated); Study Completion 2028-08-10 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Two years
  PFS was measured from the date of randomization to the date of disease progression as defined by Response Evaluation Criteria in Solid Tumor (RECIST) Version 1.1 or death

SECONDARY OUTCOMES:
Overall Survival | Three years
  OS was defined as the time from the date of randomization until death by any cause. Participants still alive at the time of data analysis were censored at the date of last follow-up.
Intracranial progression-free survival | Two years
  iPFS was defined as the time from the start of randomization to the occurrence of intracranial disease progression or death. If the subject first experiences extracranial disease progression (without concurrent intracranial disease progression), the date of first extracranial disease progression will be used as the cut-off date. For patients who have not progressed at the time of analysis, the date of their last contact will be used as the cut-off date.
Health-related quality of life per QLQ-C30 | Two years
  Health-related quality of life was evaluated using the QLQ-C30 questionnaires to assess health-related quality of life.
Health-related quality of life per QLQ-LC13 | Two years
  Health-related quality of life was evaluated using the QLQ-LC13 questionnaires to assess health-related quality of life.
Percentage of Participants With Adverse Events | Two years
  Treatment-related adverse events were assessed and graded according to CTCAE v. 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Zhengfei Zhu, MD, Principal Investigator — Fudan University; Xuwei Cai, Principal Investigator — Shanghai Chest Hospital; Qian Chu, Principal Investigator — Tongji Hospital; Xiaorong Dong, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology; Lin Wu, Principal Investigator — Hunan Cancer Hospital; Rongrong Zhou, Principal Investigator — Xiangya Hospital of Central South University; Guang Han, Principal Investigator — Hubei Cancer Hospital; Hui Zhu, Principal Investigator — Shandong Cancer Hospital and Institute; Jinjun Ye, Principal Investigator — Jiangsu Cancer Institute & Hospital; Xiaojia Cui, Principal Investigator — The Affiliated Tumor Hospital of Nantong University, Nantong, Jiangsu Province, China; Guomei Tai, Principal Investigator — The Affiliated Tumor Hospital of Nantong University, Nantong, Jiangsu Province, China; Zhiyong Yuan, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital; Dejun XIng, Principal Investigator — Jilin Provincial Tumor Hospital; Jichen Ren, Principal Investigator — Jilin Provincial Tumor Hospital; Jiancheng Li, Principal Investigator — Fujian Cancer Hospital; Yanyang Wang, Principal Investigator — General Hospital of Ningxia Medical University; Chuangzhou Rao, Principal Investigator — Ningbo No.2 Hospital; Bing Lu, Principal Investigator — The Affiliated Hospital Of Guizhou Medical University; Zhongyi Dong, Principal Investigator — Nanfang Hospital, Southern Medical University; Jiwei Liu, Principal Investigator — The First Affiliated Hospital of Dalian Medical University; Zhenzhou Yang, Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University; Hongqing Zhuang, Principal Investigator — Peking University Third Hospital; Anwen Liu, Principal Investigator — Nanchang University Second Affiliated Hospital; Haihua Yang, Principal Investigator — Taizhou Hospital Affiliated to Wenzhou Medical University; Fang Liu, Principal Investigator — Chinese PLA General Hospital; Yong Mao, Principal Investigator — Affiliated Hospital of Jiangnan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No